CLINICAL TRIAL: NCT03961932
Title: Evaluation of the Safety and Pharmacokinetics of a Single Dose of Linzagolix in Female Subjects With Normal and Impaired Renal Function
Brief Title: Safety and Pharmacokinetics of Linzagolix in Female Subjects With Normal and Impaired Renal Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ObsEva SA (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 18-OBE2109-010
Record Dates: First submitted 2019-05-20; First posted 2019-05-23 (Actual); Last update posted 2020-03-05 (Actual); Status verified 2020-03

CONDITIONS: Renal Impairment; Healthy Participants
Keywords: Linzagolix; OBE2109; Renal impairment; Renal Insufficiency; Kidney Diseases; Clinical pharmacology study
MeSH Terms: conditions — Renal Insufficiency; Kidney Diseases | interventions — linzagolix

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Normal Renal Function (Experimental): Healthy participants with Normal Renal Function (estimated Glomerular Filtration Rate (eGFR) ≥ 90 mL/min/1.73m^2)
  Interventions: Drug: Linzagolix
- Mild Renal Impairment (Experimental): Presence of Mild Renal Impairment (eGFR 60-89 mL/min/1.73m^2)
  Interventions: Drug: Linzagolix
- Moderate Renal Impairment (Experimental): Presence of Moderate Renal Impairment (eGFR 30-59 mL/min/1.73m^2)
  Interventions: Drug: Linzagolix
- Severe Renal Impairment (Experimental): Presence of Severe Renal Impairment (eGFR ≤ 29 mL/min/1.73m^2), not on hemodialysis
  Interventions: Drug: Linzagolix
- End-Stage Renal Disease (Experimental): Presence of End-Stage Renal Disease (ESRD) requiring hemodialysis
  Interventions: Drug: Linzagolix

INTERVENTIONS:
Drug: Linzagolix — A single dose of 200 mg linzagolix (2 tablets of 100 mg) will be administered orally under fasting conditions

SUMMARY:
The primary objective of this study is to assess the pharmacokinetics (PK) of linzagolix in subjects with varying degrees of impaired renal function compared to matched control subjects with normal renal function

DETAILED DESCRIPTION:
This is a Phase 1, non-randomized, open label, single-dose study to evaluate the effect of varying degrees of impaired renal function (i.e., mild, moderate, severe Renal Impairment (RI), and End-Stage Renal Disease (ESRD) on hemodialysis) on the PK, safety, and tolerability of linzagolix and its major metabolite, KP017.

Up to 40 adult female participants will be enrolled.

ELIGIBILITY:
Key Inclusion Criteria:

Renal Impaired Subjects

1. Adult female, ≥ 18 years of age at screening
2. Has a BMI ≥ 18.0 and ≤ 42.0 kg/m^2 and weight ≥ 40 kg, at screening
3. Aside from RI, be sufficiently healthy for study participation based upon medical history, physical examination, vital signs, electrocardiograms (ECGs), and screening clinical laboratory profiles, as deemed by the Principal Investigator (PI) or designee

   Subjects with mild, moderate, or severe RI:
4. Has estimated glomerular filtration rate (eGFR) based on Modification of Diet in Renal Disease (MDRD) equation at screening as follows:

   * Severe RI only: ≤ 29 mL/min/1.73m^2 not on hemodialysis
   * Moderate RI only: 30 - 59 mL/min/1.73m^2
   * Mild RI only: 60 - 89 mL/min/1.73m^2
5. Has a stable renal function with no clinically significant change in renal status at least 1 month prior to study drug administration and is not currently or has not been previously on hemodialysis for at least 1 year

   Subjects with ESRD:
6. Subject is maintained on a stable hemodialysis regimen at least 3 times a week for at least 3 months prior to dosing

Healthy Subjects

1. Health adult female will be matched to subjects with RI
2. Medically healthy with no clinically significant medical history, physical examination, laboratory profiles, vital signs or ECGs, as deemed by the PI or designee
3. Baseline eGFR ≥ 90 mL/min/1.73m^2 at screening, based on the MDRD equation. Actual creatinine clearance, as determined by a 24-hour urine collection, may be used in place of or in conjunction with the MDRD equation at the PI's discretion

Key Exclusion Criteria:

Renal Impaired Subjects

1. Had any major surgery within 4 weeks prior to dosing
2. Presence of functioning renal transplant
3. Has a surgical (e.g., hepatectomy, nephrectomy, digestive organ resection) or medical condition other than RI which might significantly alter the absorption, distribution, metabolism, or excretion of linzagolix and its metabolites, or which may jeopardize the subject's safety in case of participation in the study, in the opinion of the PI or designee

Healthy Subjects

1. Has any clinically significant illness, as judge by the PI or designee, within 4 weeks prior to dosing
2. Has laboratory values at screening or check-in which are deemed to be clinically significant (especially derangement within liver function test), unless agreed in advance by the PI and the Sponsor

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2020-01-22 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Plasma pharmacokinetic (PK) parameter Cmax of linzagolix and of KP017 | predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120 hours post-dose
  Measurement of effect of renal impairment on PK of linzagolix and its metabolite KP017 by assessment of the maximum plasma concentration (Cmax). Cmax directly determined from the plasma concentration-time profiles
Plasma PK parameter Tmax of linzagolix and of KP017 | predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120 hours post-dose
  Measurement of effect of renal impairment on PK of linzagolix and its metabolite KP017 by assessment of the Time to reach Cmax (Tmax)
Plasma PK parameter AUC0-t of linzagolix and of KP017 | predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120 hours post-dose
  Measurement of effect of renal impairment on PK of linzagolix and its metabolite KP017 by assessment of the AUC0-t (area under the concentration time curve, from time 0 to the last observed non-zero concentration)
Plasma PK parameter T1/2 of linzagolix and of KP017 | predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120 hours post-dose
  Measurement of effect of renal impairment on PK of linzagolix and its metabolite KP017 by assessment of the T1/2 (Terminal half life)

SECONDARY OUTCOMES:
Treatment emergent Adverse Events | Day 1 to 14 days post-dose
  Assessment of safety and tolerability of a single dose linzagolix in renal impaired subjects compared with healthy control subjects by assessing the number, frequency and severity of treatment emergent Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: ObsEva SA, Study Director — Geneva
Locations (2):
- United States (2):
  - Clinical Site, Orlando, Florida
  - Clinical Site, Saint Paul, Minnesota